CLINICAL TRIAL: NCT02166567
Title: The Effect of Sorting of Non-apoptotic and Apoptotic Spermatozoa Using Flow Cytometry on the Outcome of Intracytoplasmic Sperm Injection.
Brief Title: Effect of Sorting of Apoptotic Spermatozoa on the Outcome of Assisted Reproduction
Acronym: Spermsorting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EKBB178/12; YOPRO (Other: University of Basel)
Record Dates: First submitted 2014-06-14; First posted 2014-06-18 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Male Infertility
Keywords: intracytoplasmic sperm injection; Male infertility; apoptosis; flow cytometry and sorting; DNA fragmentation
MeSH Terms: conditions — Infertility, Male | interventions — Flow Cytometry

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YoPro and FACS (Experimental): Spermatozoa to be used for ICSI will be stained with the YoPro Dye and then be sorted with FACS to select non-YoPro stained spermatozoa, known to have significantly less fragmented DNA.
  Interventions: Procedure: Staining of spermatozoa with the YoPro dye and sorting of the stained spermatozoa with FACS
- Swim-up (Active Comparator): Spermatozoa will be processed using the conventional swim-up me
  Interventions: Procedure: Swim-up

INTERVENTIONS:
Procedure: Staining of spermatozoa with the YoPro dye and sorting of the stained spermatozoa with FACS
  Other Names: YoPro; FACS
  Arms: YoPro and FACS
Procedure: Swim-up — Semen processing will be carried out with the conventional swim-up method.
  Arms: Swim-up

SUMMARY:
In assisted reproductive technology (ART) semen needs to be processed. Commonly used methods rely on physical properties of the spermatozoa, such as the swim-up methods and density gradient centrifugation. It is now known that current processing of spermatozoa does not prevent the admixture of spermatozoa with damaged genetic material. The latter have a negative impact on the outcome of ART. The investigators developed a new method for the processing of spermatozoa with intact genetic material based on flow cytometry and sorting (FACS) and on staining using a deye, YoPro. The investigators aim at examining the effect of this novel method of sperm sorting on the outcome of ART.

ELIGIBILITY:
Inclusion Criteria:

* infertile couples needing treatment with ICSI
* male infertility as defined by the WHO 2010 criteria
* age of the treated women should be between 22 and 39 years of age.
* normal ovarian reserve, as defined by basal FSH-concentration below 10 IU/l and AMH-concentration above 10 pmol/l.
* signed consent form.

Exclusion Criteria:

* normal male infertility, as defined by the WHO 2010 criteria
* age of the treated women below 22 years and above 39 years
* reduced ovarian reserve, as defined by an elevated basal FSH-concentration or reduced AMH-concentration.
* Not more than two preceding unsuccessfull treatments with ICSI
* Severe disease of the male or female partner, such as HIV, hepatitis, or psychiatric illness.
* Participation in another study.
* lack of a signed consent form.

Ages: 22 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2017-01 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | Week 12 of gestation

SECONDARY OUTCOMES:
Number of diploidic fertilized oocytes. | one day after intracytoplasmic sperm injection

OTHER OUTCOMES:
Number of embryos growing to the blastocyst stage | 5 days after intracytoplasmic sperm injection
Implantation rate, e.g. number of implanted embryos with heart activity per number of embryos transferred | week 12 of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Geyter, MD, Prof., Principal Investigator — Univeristy Hospital Basel
Locations (1):
- University of Basel, Basel, Basel BS, Switzerland

REFERENCES:
- [Background] Ribeiro SC, Sartorius G, Pletscher F, de Geyter M, Zhang H, de Geyter C. Isolation of spermatozoa with low levels of fragmented DNA with the use of flow cytometry and sorting. Fertil Steril. 2013 Sep;100(3):686-94. doi: 10.1016/j.fertnstert.2013.05.030. Epub 2013 Jun 27. PMID 23809499
- [Derived] De Geyter C, Gobrecht-Keller U, Ahler A, Fischer M. Removal of DNA-fragmented spermatozoa using flow cytometry and sorting does not improve the outcome of intracytoplasmic sperm injection. J Assist Reprod Genet. 2019 Oct;36(10):2079-2086. doi: 10.1007/s10815-019-01571-1. Epub 2019 Aug 28. PMID 31463874